CLINICAL TRIAL: NCT06580275
Title: The GLACE Study: A Prospective Multi-center Single Arm Study Evaluating the Safety and Performance of the CLAAS Device With ICE Guided LAA Closure.
Brief Title: The GLACE Study: Evaluating CLAAS With ICE Guided LAA Closure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Conformal Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 24-101
Record Dates: First submitted 2024-08-26; First posted 2024-08-30 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation; Stroke Prevention
Keywords: Atrial fibrillation; Stroke; ICE; Conformal; LAAO
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- CLAAS (Experimental): In this single arm study, all eligible subjects will be assigned to receive the CLAAS device.
  Interventions: Device: CLAAS

INTERVENTIONS:
Device: CLAAS — All eligible subjects will have an LAA closure attempt using the CLAAS device guided by ICE technology.

SUMMARY:
The CLAAS® device will be evaluated for safety and performance in the reduction of stroke in subjects with non-valvular atrial fibrillation under intracardiac echocardiography (ICE) imaging for left atrial appendage closure.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female aged ≥18 years.
2. Documented non-valvular AF (paroxysmal, persistent, or permanent).
3. High risk of stroke or systemic embolism, defined as CHADS2 score of ≥2 or CHA2DS2-VASc score of ≥3.
4. Has an appropriate rationale to seek a non-pharmacologic alternative to long-term oral anticoagulation including contraindications to long term oral anti-coagulation inclusive of history of intracranial bleed, subdural hematoma, gastrointestinal bleeding, hematuria, epistaxis, falls, and other less common conditions. Also included is the inability to reliably take medications and reluctance to take a blood thinner.
5. Deemed by investigator to be suitable for short term oral anticoagulation therapy but deemed less favorable for long-term oral anticoagulation therapy.
6. Deemed appropriate for LAA closure by the site investigator and a clinician not a part of the procedural team using a shared decision-making process in accordance with standard of care.
7. Able to comply with the protocol-specified medication regimen and follow-up evaluations.
8. The patient has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent approved by the appropriate institutional review board (IRB)/Regional Ethics Board (REB)/Ethics Committee (EC).

Exclusion Criteria:

1. Pregnant or nursing patients and those who plan pregnancy in the period up to one year following the index procedure. Female patients of childbearing potential must have a negative pregnancy test (per site standard test) within 7 days prior to index procedure.
2. Anatomic conditions that would prevent performance of an LAA occlusion procedure (e.g., prior atrial septal defect [ASD] or patent foramen ovale [PFO], surgical repair or implanted closure device, or obliterated or ligated left atrial appendage).
3. Atrial fibrillation that is defined by a single occurrence or that is transient or reversible (e.g., secondary thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures).
4. A medical condition (other than atrial fibrillation) that mandates long-term oral anticoagulation (e.g., history of unprovoked deep vein thrombosis or pulmonary embolism, or mechanical heart valve).
5. History of bleeding diathesis or coagulopathy, or patients in whom antiplatelet and/or anticoagulant therapy is contraindicated.
6. Documented active systemic infection.
7. Symptomatic carotid artery disease (defined as >50% stenosis with symptoms of ipsilateral transient or visual TIA evidenced by amaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral stroke); if subject has a history of carotid stent or endarterectomy the subject is eligible if there is <50% stenosis noted at the site of prior treatment.
8. Recent (within 30 days of index procedure) or planned (within 60 days post-procedure) cardiac or non-cardiac interventional or surgical procedure.
9. Recent (within 30 days of index procedure) stroke or transient ischemic attack.
10. Recent (within 30 days of index procedure) myocardial infarction.
11. Vascular access precluding delivery of implant with catheter-based system.
12. Severe heart failure (New York Heart Association Class IV).
13. Prior cardiac transplant, history of mitral valve replacement or transcatheter mitral valve intervention, or any mechanical valve implant.
14. Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) <30mL/min/1.73 m2 (by the Modification of Diet in Renal Disease equation).
15. Platelet count <75,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <3,000 cells/mm3.
16. Known allergy, hypersensitivity or contraindication to aspirin, heparin, or device materials (e.g., nickel, titanium) that would preclude any P2Y12 inhibitor therapy, or the patient has contrast sensitivity that cannot be adequately pre-medicated.
17. Actively enrolled or plans to enroll in a concurrent clinical study in which the active treatment arm may confound the results of this study.
18. Unable to undergo general anesthesia.
19. Known other medical illness or known history of substance abuse that may cause non-compliance with the protocol or protocol-specified medication regimen, confound the data interpretation, or is associated with a life expectancy of less than 5 years.
20. A condition which precludes adequate transesophageal echocardiographic (TEE) assessment or ICE guided imaging during the procedure.

Imaging Exclusion Criteria:

1. Left atrial appendage anatomy which cannot accommodate the CLAAS device per manufacturer IFU (e.g., the anatomy and sizing must be appropriate for the test (CLAAS) device in order to be enrolled in the trial).
2. Intracardiac thrombus or dense spontaneous echo contrast consistent with thrombus, as visualized by pre-procedural imaging (TEE or Cardiac CT) or baseline procedural ICE prior to implant.
3. Left ventricular ejection fraction (LVEF) <30%.
4. Moderate or large circumferential pericardial effusion >10mm or symptomatic pericardial effusion, signs or symptoms of acute or chronic pericarditis, or evidence of tamponade physiology.
5. Atrial septal defect that warrants closure.
6. High risk patent foramen ovale (PFO), defined as an atrial septal aneurysm (excursion >15mm or length >15mm) or large shunt (early [within 3 beats] and/or substantial passage of bubbles, e.g., ≥20).
7. Moderate or severe mitral valve stenosis (mitral valve area <1.5cm2).
8. Complex atheroma with mobile plaque of the descending aorta and/or aortic arch.
9. Evidence of cardiac tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Successful LAA closure (Evaluated at 45 Days Post-procedure) | 45 Days
  Complete closure is defined as absence of a significant leak (>5 mm) as assessed based upon core lab evaluation of 45 Day Imaging assessment without device or procedure related SAEs.
Successful LAA closure without procedural complication within 7 days post-procedure | 7 Days
  The absences of any of the following complications: Cardiac perforation, pericardial effusion requiring drainage, ischemic stroke, device embolization, and major vascular complications.

SECONDARY OUTCOMES:
Stroke: Ischemic, Hemorrhagic, Disabling, Non-Disabling | 12 Months
Bleeding (BARC 3-5) | 14 Days
  Procedural and Non-Procedural
Device Leak | 45 Days
  >5 mm, 3-5 mm, 1-3 mm leak is based on core lab imaging assessment at 45 days
Pericardial Effusion requiring drainage | 12 Months
Procedural and Device related AEs and SAEs | 1 Day
Device Success | 1 Day
  CLAAS implantation in correct position without complications till discharge
Conversion to TEE | 1 Day
Conversion to general anesthesia (GA) with endotracheal intubation | 1 Day

CONTACTS AND LOCATIONS:
Locations (4):
- Na Homolce Hospital, Prague, Czechia
- Denmark (2):
  - Aarhus University Hospital, Skejby, Aarhus
  - University Hospital of Copenhagen, Copenhagen
- Fondazione Toscana Gabriele Monasterio, Massa, Italy